CLINICAL TRIAL: NCT03265743
Title: HPV (Papilloma Human Virus) Vaccination in Young Women With Cystic Fibrosis and Followed in the Auvergne Rhône-Alpes Region
Brief Title: HPV Vaccination in Women With Cystic Fibrosis
Acronym: VACCIN-HPV-MUC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0277
Record Dates: First submitted 2017-07-27; First posted 2017-08-29 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-07

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Cystic Fibrosis: Patients with Cystic Fibrosis, followed in a pediatric or mixed Cystic Fibrosis center of the region Auvergne Rhône Alpes (AuRA), aged 11 years or older.
  Interventions: Other: Self-report Written Questionnaire

INTERVENTIONS:
Other: Self-report Written Questionnaire — Informations are gathered through a self-report written questionnaire, completed by the patients or their parents.

SUMMARY:
The main risk factor for the development of cervical lesions is human papillomavirus (HPV) infection. Vaccination against human papillomavirus, which is offered to all girls aged 11 to 14, and catching up to girls aged 15 to 19, is an effective method of preventing cervical pathology. Despite this, human papillomavirus vaccination coverage remains low in France.

Some women with cystic fibrosis might need a transplantation, which is a factor associated with increased risk of human papillomavirus carriage and cervical pathology. An over-risk of cervical pathology would also be present in non-transplanted women with cystic fibrosis. Particular attention should therefore be paid to vaccination in this population.

The objective is to estimate the frequency of human papillomavirus vaccination in young patients with cystic fibrosis, and to evaluate the reasons for non-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* girls with Cystic Fibrosis
* followed in a pediatric or mixed Cystic Fibrosis center of the region Auvergne Rhône Alpes (AuRA)
* aged 11 years or older

Exclusion Criteria:

- Refusal to respond to the questionnaire

Ages: 11 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Study Population: This study is intended for girls with Cystic Fibrosis, followed in a pediatric or mixed Cystic Fibrosis center of the region Auvergne Rhône Alpes (AuRA), aged 11 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Realization of human papillomavirus vaccination | 15 minutes
  The main outcome is the prevalence of human papillomavirus vaccination in young women with Cystic fibrosis.
  This data is collected using a questionnaire : HPV vaccination performed : yes/no

SECONDARY OUTCOMES:
Type of vaccine used | 15 minutes
  This data is collected using a questionnaire : bivalent (Cervarix®) or quadrivalent (Gardasil®)
Respect for the vaccinal plan | 15 minutes
  This data is collected using a questionnaire : number and dates of injections
Reasons for non-vaccination | 15 minutes
  In case of non-vaccination reasons are collected using a multiple choices questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Nouvel Hôpital d'Estaing CRCM Mixte, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Cystic Fibrosis Reference Center, Hospices Civils de Lyon, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No